CLINICAL TRIAL: NCT02572908
Title: Effects of Wheat Breads on Symptoms of IBS, a Pilot Study
Acronym: Wheat-IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oy Karl Fazer Ab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Wheat-IBS
Record Dates: First submitted 2015-10-05; First posted 2015-10-09 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Irritable Bowel Syndrome; Wheat Sensitivity
Keywords: wheat, IBS, gluten, ATI
MeSH Terms: conditions — Irritable Bowel Syndrome; Ichthyosis Bullosa of Siemens | interventions — Diet, Gluten-Free

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Fermented wheat bread for 7 days (Active Comparator): Long sourdough fermentation
  Interventions: Other: Sourdough wheat bread; Other: Gluten-free diet
- Yeast baked wheat bread for 7 days (Placebo Comparator): Regular toast bread
  Interventions: Other: Regular yeast baked toast bread; Other: Gluten-free diet
- Run-in (Other): Gluten-free diet for 7 days before entering either bread period
  Interventions: Other: Gluten-free diet

INTERVENTIONS:
Other: Sourdough wheat bread
  Arms: Fermented wheat bread for 7 days
Other: Regular yeast baked toast bread
  Arms: Yeast baked wheat bread for 7 days
Other: Gluten-free diet — Gluten-free diet excluding even oats and buckwheat. Rice, quinoa, corn and potato allowed as grains/pseudo-grains

SUMMARY:
This is randomized pilot study comparing tolerability of yeast-baked wheat bread and sourdough wheat bread in irritable bowel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* IBS & subjective sensitivity to wheat

Exclusion Criteria:

* celiac disease, pregnancy, lactation, IBD, major GI operations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Subjective symptoms using visual analog scale (VAS) daily | 7 days
  Self-reports of bloating, dyspepsia, constipation, diarrhoea, abdominal pain, borborygmi, flatulence, heart burn, urgency to defecate, incomplete feeling of defecation, abdominal cramps, tiredness, skin rash, mood, nausea, joint pain, ability to concentrate and loss of appetite on VAS 0-100. Participants fill in VAS questionnaires at the end of each day

CONTACTS AND LOCATIONS:
Locations (1):
- Aava Medical Centre, Helsinki, Helsinki, Finland